CLINICAL TRIAL: NCT00134576
Title: Automated Assessment of Mental Health in the Workplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Dr. Ramesh Farzanfar, Boston University
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: R01DP000116 (NIH)
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-05

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Computer Assisted Education for Behavioral Change — TLC-Detect will provide subjects in the intervention group with information about each diagnosed mental health disorder. TLC-Detect will then give the Treatment Module and will tell the intervention subjects that it will call back in one month for a follow-up or the next week if a subject is comorbid with other disorders.

SUMMARY:
The purpose of this study is to design, refine, and test for the effectiveness of a computer-based telephone system (Telephone-Linked Communications for Detection of Mental Health Disorders in the Workplace; TLC-Detect) that will screen workers for mental health distress; educate them about seeking treatment; and follow up with them over a 6 month period.

ELIGIBILITY:
Inclusion Criteria:

* Employment with benefits at Boston Medical Center, Boston University, or Florida Power and Light Company
* Ability to speak and understand conversational English
* > 18 years of age
* Access to a touch-tone telephone
* Screen positive for the World Health Organization (WHO)-5 Well-Being Index

Exclusion Criteria:

* Being under treatment (medication or therapy) for a mental health disorder
* Taking medication for a serious/major medical disorder that interferes with normal life
* Taking medication prescribed for mental health treatment on a daily basis
* Diagnosed with schizophrenia
* Planning to go on leave for over 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Absenteeism and presentism (functionality at work), measured every three months for 6 months | 6 months

SECONDARY OUTCOMES:
Treatment status, timing of measurement depends upon symptom severity | 6 months
Health status measured every three months for 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Farzanfar, PhD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States